CLINICAL TRIAL: NCT04011709
Title: An Open-label, Non-drug Methodology Trial to Evaluate the Use of a Mouthpiece With the VR647 Inhalation System During Delivery of Isotonic Saline (0.9% NaCl) in Subjects Less Than Five Years of Age Who Have Previously Received an Inhaled Therapy Delivered Either by a Nebulizer or by a Pressurized Metered-dose Inhaler Plus Spacer
Brief Title: A Methodology Trial Using the VR647 Inhalation System in Pediatric Subjects Who Have Previously Received Inhaled Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vectura Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR647/0/003
Record Dates: First submitted 2019-06-17; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Cough; Wheezing
Keywords: Nebulizer; Pediatric; Methodological study
MeSH Terms: conditions — Cough; Respiratory Sounds

STUDY DESIGN:
Intervention Model Description: This open-label, non-drug methodology trial consists of a screening assessment, familiarization session and a nebulization assessment at one visit and a second nebulization assessment at a second visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Visit 1 and Visit 2, Test Arm 2A (Other): Subjects who carried out 3 attempts at Visit 1, failed to achieve nebulization success and subsequently were included in Test Arm 2A for Visit 2
  Interventions: Combination Product: VR647 Inhalation System + VR647 Smart Card 3 Secs; Combination Product: VR647 Inhalation System + VR647 Smart Card 2 Secs
- Visit 1 and Visit 2, Test Arm 2B (Other): Subjects who carried out 3 attempts at Visit 1, achieved nebulization success and were subsequently included in Test Arm 2B for Visit 2
  Interventions: Combination Product: VR647 Inhalation System + VR647 Smart Card 3 Secs; Combination Product: VR647 Inhalation System + VR647 Smart Card 4 Secs

INTERVENTIONS:
Combination Product: VR647 Inhalation System + VR647 Smart Card 3 Secs — 3 attempts of 19 inhalations, 3 second per breath. Attempts 1 and 2 will be made with air only. Attempt 3 will be made with isotonic saline (0.9% NaCl)
Combination Product: VR647 Inhalation System + VR647 Smart Card 2 Secs — 3 attempts of 28 inhalations, 2 second per breath. Attempts 1 and 2 will be made with air only. Attempt 3 will be made with isotonic saline (0.9% NaCl)
  Arms: Visit 1 and Visit 2, Test Arm 2A
Combination Product: VR647 Inhalation System + VR647 Smart Card 4 Secs — 3 attempts of 14 inhalations, 4 second per breath. Attempts 1 and 2 will be made with air only. Attempt 3 will be made with isotonic saline (0.9% NaCl)
  Arms: Visit 1 and Visit 2, Test Arm 2B

SUMMARY:
This is an open-label, non-drug methodology trial in which subjects undergo a stepwise series of tests to evaluate their ability to use a mouthpiece to deliver nebulized therapy.

The trial consists of a screening assessment and familiarization session, and two nebulization assessments, conducted over two site visits. The screening assessment, familiarization session and first nebulization assessment will take place at Visit 1, while the second nebulization assessment will take place at Visit 2. The total duration between Visits 1 and 2 will be 4 - 8 days. Each visit is expected to last up to 2 hours.

DETAILED DESCRIPTION:
At the initial visit (Visit 1), eligible subjects (i.e., children) and their parent(s)/legal guardian(s) will be approached to ascertain their interest in trial participation. Interested subjects and their parent(s)/legal guardian(s) will proceed to a nebulizer familiarization session. After informed consent has been obtained from the subject's parent(s)/legal guardian(s), the subject will proceed to Nebulization Assessment 1.

At Nebulization Assessment 1 (Visit 1), all subjects will perform 3 attempts of 19 inhalations, each inhalation of 3 seconds duration. Nebulization Assessment 2 (Visit 2) will occur 4-8 days after Visit 1. Subjects, who failed to achieve nebulization success at Attempt 3 during Visit 1, will perform 3 attempts of 28 inhalations, each inhalation of 2 seconds duration at Visit 2. Subjects, who achieved nebulization success at Attempt 3 during Visit 1, will perform 3 attempts of 14 inhalations, each inhalation of 4 seconds duration at Visit 2.

At each visit, Attempts 1 and 2 will be made with air only. Attempt 3 will be made with isotonic saline (0.9% NaCl). Nebulization success will be assessed at Attempt 3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 1 to <5 years
* History of coughing and/or recurrent wheezing within the last year, otherwise healthy
* Use of an inhaler with a spacer or nebulizer for at least 30 days (consecutive or otherwise) within the last year. Examples of inhaled or nebulized therapy include the use of a regular controller (inhaled corticosteroids (ICS) or ICS/long-acting beta-agonists), or a reliever therapy (e.g., albuterol) on an as needed basis for the relief of symptoms
* Written informed consent from the subjects's parent(s)/legal guardian(s), including privacy authorization, prior to trial participation
* Subject's parent(s)/legal guardian(s) must be willing and able to comply with the trial procedures and visit schedules

Exclusion Criteria:

Screening (Visit 1)

* Any significant medical conditions (apart from a history of coughing and/or recurrent wheezing) that in the opinion of the investigator would interfere with the subject's ability to use the mouthpiece and/or follow the protocol procedures
* Subjects with current respiratory symptoms or breathing difficulties at the time of screening
* History of paradoxical bronchospasm or hyper-responsiveness following inhaled therapy that in the opinion of investigator may put the subject at risk when inhaling isotonic saline
* Parent(s)/legal guardian(s) who is an employee of the investigational site or the Sponsor, who is directly involved in the trial, or a family member of such a person

Nebulization Assessment 2 (Visit 2)

* Development of any new illness or condition between the Screening (Visit 1) and prior to Nebulization Assessment 2 (Visit 2) that in the opinion of the investigator would interfere with the subject's ability to use the mouthpiece and/or follow the protocol procedures
* Any safety concerns that in the opinion of the investigator would jeopardize the subject by his/her continued participation in the trial

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects achieving nebulization success using a mouthpiece overall and by age (years) at each visit. | 4 to 8 days
  Nebulization success using a mouthpiece defined as actuating the nebulizer on at least 70% of planned inhalations and inhaling at least 50% of the total intended inhalation volume.

SECONDARY OUTCOMES:
Number of breaths completed by subjects using a mouthpiece overall and by age (years) at each visit. | 4 to 8 days
  Number of breaths completed by subjects using a mouthpiece recorded at each visit.
Number of subjects aged 3 to <5 years who require parent(s)/legal guardian(s) hands-on assistance at Attempt 3 at each visit. | 4 to 8 days
  Number of subjects aged 3 to <5 years who require parent(s)/legal guardian(s) hands-on assistance as assessed (Yes/No) by the Investigator on the inhalation checklist.
Number of subjects who require parent(s)/legal guardian(s) hands-on assistance at Attempt 3 overall and by age (years) at each visit. | 4 to 8 days
  Number of subjects who require parent(s)/legal guardian(s) hands-on assistance as assessed (Yes/No) by the Investigator on the inhalation checklist.
The quality of nebulization at Attempt 3 as recorded in the inhalation checklist overall and by age (years) at each visit. | 4 to 8 days
  The inhalation checklist consists of 5 questions regarding inhalation quality answered Yes/No (Q1, Q2, Q3 and Q5) or by percentage (Q4), with Yes answers for Q1-3 and >50% for Q4 (or Yes answers for Q1-3 and Q5 in the successful subgroup analysis) being scored as perfect.
Mean modified Patient Satisfaction and Preference Questionnaire (PASAPQ) total score at Attempt 3 at Visit 2 overall and by age (years). | 4 to 8 days
  The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices. The modified PASAPQ consists of 10 questions. The first 8 questions generate the total score domain (scale: 1 (i.e., very dissatisfied) to 7 (i.e., very satisfied); range: 14.3 to 100, calculated as ((Q1+Q2+Q3+Q4+Q5+Q6+Q7+Q8)/56)*100).
Mean modified PASAPQ satisfaction score at Attempt 3 at Visit 2 overall and by age (years). | 4 to 8 days
  The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices. The modified PASAPQ consists of 10 questions. Question 9 asks for overall satisfaction with the device(s) used in the trial (scale: 1 (i.e., very dissatisfied) to 7 (i.e., very satisfied); range: 1-7).
Mean modified PASAPQ score indicating willingness to continue with the device at Attempt 3 at Visit 2 overall and by age (years). | 4 to 8 days
  The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices. The modified PASAPQ consists of 10 questions. Question 10 asks about willingness to continue with the device(s) used in the trial (scale: 0 (i.e, not willing) to 100 (i.e., definitely willing; range: 0-100).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Burgess, MD, Study Director — Vectura Ltd
Locations (5):
- United States (5):
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Clinical Research Institute, Inc, Plymouth, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - North Carolina Clinical Research, Raleigh, North Carolina
  - National Allergy and Asthma Research, LLC, Charleston, South Carolina